CLINICAL TRIAL: NCT03727932
Title: VioOne™ HIV Profile™ Supplemental Assay
Brief Title: VioOne HIV Profile Supplemental Assay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avioq, Inc. (Industry)
Collaborators: Clinical Reference Laboratory (Industry); Duke Clinical Research Institute (Other); University of North Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 100004
Record Dates: First submitted 2018-10-25; First posted 2018-11-01 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-11

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- VioOne HIV Profile (Other): HIV Profile™ is intended as an aid in the diagnosis of infection with HIV-1 and/or HIV-2. It is intended as an additional, more specific test to confirm the presence of antibodies to HIV-1 and HIV-2 for specimens repeatedly reactive in diagnosis or screening procedures, including pediatric patients (ages 2-20).
  Interventions: Device: VioOne HIV Profile Supplemental Assay

INTERVENTIONS:
Device: VioOne HIV Profile Supplemental Assay — The VioOne™ HIV Profile™ Supplemental Assay is an enzyme-linked immunosorbent assay (ELISA) for confirmation and differentiation of individual antibodies directed to various gene products of Human Immunodeficiency Virus Type 1 (HIV-1 Group M & Group O) and Type 2 (HIV-2) in human serum or plasma. The HIV Profile™ is intended as an aid in the diagnosis of infection with HIV-1 and/or HIV-2.

SUMMARY:
Assessment of the sensitivity, specificity and reproducibility of the VioOne HIV Profile Supplemental Assay

DETAILED DESCRIPTION:
Specificity A total of 280 serum samples and 300 plasma samples from a low-risk population (e.g. blood donors) will be collected at Houston Gulf Coast Regional Blood Center (Houston, TX). All serum and plasma specimens will be previously screened and found non-reactive with FDA licensed or approved HIV-1/2 assays (a population of samples that would not normally be tested with the Avioq VioOne™ HIV Profile™ Supplemental Assay). The number of serum samples will be supplemented up to 300 with the inclusion of 20 pediatric samples; 10 from children aged 2 - 11 and 10 from children aged 12-18 for a total of 600 samples for specificity testing. Samples will be tested with one of three validation kit lots of the Avioq VioOne TM HIV Profile™ Supplemental Assay manufactured at Avioq.

The samples will be tested at 3 external sites in proportions based on the manufacturing size of the individual validation lots. At Site 1 the samples will be further divided approximately 70% I 30% between Validation lots 1 & 2. At Site 2 the samples will be divided approximately 70% / 30%, between Validation lots 2 and 3. At site 3 the samples will be tested entirely with Validation lot 3. The study design calls for the use of at least one lot in common at all 3 clinical sites based on a request from the FDA.

For the Specificity Study, any indeterminate or reactive samples will be tested with either the FDA approved Bio-Rad Geenius assay or Western Blot to determine the true classification. Specificity and 95% confidence intervals will be calculated.

Sensitivity Serum or plasma (n= 757) repository samples from individuals infected with HIV will be tested at four external sites and at Avioq with up to four validation kit lots. The samples will be tested at all sites in proportions based on the manufacturing size of the individual validation lots. At Site 1 the samples will be further divided approximately 75% I 25% between Validation lots 1 & 2. At Site 2 the samples will be divided approximately 75% / 25%, between Validation lots 2 and 3. At sites 3 and 4 the samples will be tested entirely with Validation lot 3. A fourth lot (Validation lot 5) will be used to test a few HIV-1 Group O samples at Avioq. The study design calls for the use of at least one lot in common at all 4 clinical sites based on a request from the FDA.

The sensitivity samples will consist of 400 HIV positives, a minimum of 200 HIV-2 positives, 50 AIDS positive, 40 pediatric HIV positive, a minimum of 15 HIV-O positives, 10 HIV-1/HIV-2 coinfected positives and a minimum of 27 samples from pregnant females (samples from all three trimesters) infected with HIV.

All specimens are expected to be positive for HIV-1 and/or HIV-2 antibody representing the types of specimens expected to be tested with the Avioq VioOne™ HIV Profile™ Supplemental Assay. Samples with VioOne™ HIV Profile™ assay results discordant from this expectation will be resolved by testing the same samples in FDA approved confirmatory assays such as the BioRad Geenius or Western Blot.

ELIGIBILITY:
Inclusion Criteria:

* Specificity = 280 Serum Samples and 300 Plasma Samples
* An additional 20 Serum pediatric samples
* From low risk population (e.g. blood donors)
* Sensitivity = 757 Total Samples

  * 400 HIV positive,
  * 200 HIV-2 positive
  * 50 AIDS positive
  * 40 Pediatric
  * 15 HIV-O positive
  * 10 HIV-1/HIV-2 co-infected positive
  * 27 samples from pregnant females with HIV

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 757 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2018-04-11 (Actual); Study Completion 2018-04-11 (Actual)

PRIMARY OUTCOMES:
Clinical specificity and sensitivity of HIV Infection | 9 months
  Clinical Specificity and 95% CI of the Profile Assay Clinical Sensitivity and 95% CI of the Profile Assay

CONTACTS AND LOCATIONS:
Locations (1):
- Avioq Inc, Research Triangle Park, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No